CLINICAL TRIAL: NCT03393091
Title: Perioperative Anaphylaxis in Patients Attending University Hospitals (Egypt - United Kingdom).
Brief Title: Perioperative Anaphylaxis in Patients Attending University Hospitals (Egypt - UK).
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hytham Hussien Kamel Mohamed Shoeib, Principal investigator, Assiut University
Other Study IDs: AssiutU222
Record Dates: First submitted 2017-12-28; First posted 2018-01-08 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Perioperative/Postoperative Complications; Drug-Induced Anaphylaxis
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Incidence of possible anaphylaxis: Data will be collected on 1000 consecutive general anaesthetic procedures in Assiut University Hospitals. After each elective operating list the anaesthetist will be asked to complete a form in which they will document the number of patients receiving general anaesthesia on the list and the number of those patients who developed any of the following features: unexpected, unexplained hypotension; unexpected bronchospasm resistant to treatment; angioedema; urticaria; severe itching; widespread erythema

SUMMARY:
Perioperative anaphylaxis is associated with significant morbidity and mortality. Most textbooks describe it as a rare event of the order of 1 in 10 to 1 in 20,000 general anaesthetic cases. However, a recent study in the United Kingdom suggested that 1 in 350 cases have features suspicious of perioperative anaphylaxis. This study suggests that perioperative anaphylaxis may be under recognised and under reported.

When perioperative anaphylaxis is recognised, it would be ideal to carry out investigations firstly to confirm the diagnosis of anaphylaxis and secondly to identify the causative agent. The latter can be difficult in the context of anaesthesia where the patient is exposed to several drugs and other reagents in a short space of time.

One of the interesting aspects of perioperative anaphylaxis is that there is variability in its epidemiology between different countries, for example between the United Kingdom, France, Scandinavia and Australia and New Zealand. There are currently no data from Egypt to include in such comparisons and to inform clinical practice.

As well as being at risk if a drug allergen is not identified, patients can also be at risk from an incorrect allergy label. The most common example of this is penicillin allergy where fewer than 10% of patients with a history of penicillin allergy are found to be allergic. Incorrect penicillin allergy labels are potentially harmful for patients attending for surgery because the label independently increases the risk of developing infection to resistant organisms, longer hospital stays and mortality.

DETAILED DESCRIPTION:
Perioperative anaphylaxis is associated with significant morbidity and mortality. Most textbooks describe it as a rare event of the order of 1 in 10 to 1 in 20,000 general anaesthetic cases. However, a recent study in the United Kingdom suggested that 1 in 350 cases have features suspicious of perioperative anaphylaxis. This study suggests that perioperative anaphylaxis may be under recognised and under reported.

When perioperative anaphylaxis is recognised, it would be ideal to carry out investigations firstly to confirm the diagnosis of anaphylaxis and secondly to identify the causative agent. The latter can be difficult in the context of anaesthesia where the patient is exposed to several drugs and other reagents in a short space of time.

One of the interesting aspects of perioperative anaphylaxis is that there is variability in its epidemiology between different countries, for example between the United Kingdom, France, Scandinavia and Australia and New Zealand. There are currently no data from Egypt to include in such comparisons and to inform clinical practice.

As well as being at risk if a drug allergen is not identified, patients can also be at risk from an incorrect allergy label. The most common example of this is penicillin allergy where fewer than 10% of patients with a history of penicillin allergy are found to be allergic. Incorrect penicillin allergy labels are potentially harmful for patients attending for surgery because the label independently increases the risk of developing infection to resistant organisms, longer hospital stays and mortality.

Aim of the work:

This project proposes the following studies:

1. The incidence of suspected perioperative anaphylaxis in an Egyptian population.
2. Sensitivity and specificity of tryptase changes under surgery and anaesthesia.

Patient and Methods:

1. In order to define the incidence of possible anaphylaxis, data will be collected on 1000 consecutive general anaesthetic procedures in Assiut University Hospitals. After each elective operating list the anaesthetist will be asked to complete a form in which they will document the number of patients receiving general anaesthesia on the list and the number of those patients who developed any of the following features: unexpected, unexplained hypotension; unexpected bronchospasm resistant to treatment; angioedema; urticaria; severe itching; widespread erythema.
2. Tryptase is a relatively stable protein released from mast cells alongside histamine during allergic anaphylaxis. Mast cell tryptase is recognised as a useful biomarker for perioperative anaphylaxis but there is debate concerning what degree of change in mast cell tryptase produces the greatest combination of sensitivity and specificity for perioperative anaphylaxis. Variable results from different countries suggest that population specific normal responses may need to be defined.

This study will be conducted in Assiut University Hospitals. A blood cell sample for mast cell tryptase will be taken immediately prior to surgery and 1 hour following induction of anaesthesia in the following groups of patients (n = 30 in each case):

1. Children undergoing elective surgery between the ages of 3 and 10 years
2. Adults between the ages of 16 and 30 years undergoing orthopaedic trauma surgery
3. Adults more than 60 years of age undergoing orthopaedic surgery
4. Women of any age undergoing gynaecological surgery
5. Adults of any age undergoing emergency general surgery
6. Adults undergoing cardiac surgery involving cardiopulmonary bypass (samples will be taken immediately preoperatively, prior to cardiopulmonary bypass and 1 hour after cardiopulmonary bypass)
7. Women undergoing caesarean section under general or regional anaesthesia

ELIGIBILITY:
Inclusion Criteria:

* In order to define the incidence of possible anaphylaxis, data will be collected on 1000 consecutive general anaesthetic procedures in Assiut University Hospitals.
* A blood cell sample for mast cell tryptase will be taken immediately prior to surgery and 1 hour following induction of anaesthesia in the following groups of patients (n = 30 in each case):

  (a) Children undergoing elective surgery between the ages of 3 and 10 years (b) Adults between the ages of 16 and 30 years undergoing orthopaedic trauma surgery (c) Adults more than 60 years of age undergoing orthopaedic surgery (d) Women of any age undergoing gynaecological surgery (e) Adults of any age undergoing emergency general surgery (g) Women undergoing caesarean section under general or regional anaesthesia

Exclusion criteria:

patient refusal, history of previous allergic reaction.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Data will be collected on 1000 consecutive general anaesthetic procedures in Assiut University Hospitals.
  * A blood cell sample for mast cell tryptase will be taken immediately prior to surgery and 1 hour following induction of anaesthesia in the previously mentioned groups of patients (n = 30).
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of suspected perioperative anaphylaxis in an Egyptian population. | one year
  Snap shot on epidemiology of perioperative hypersensitivity reactions in an Egyptian population

SECONDARY OUTCOMES:
Effect of anaesthesia and surgery on mast cell tryptase | two years
  Study effect of age, sex, anaesthesia, fluid and surgery on mast cell tryptase in control and reaction groups

CONTACTS AND LOCATIONS:
Overall Officials: Hytham Shoeib, MCs,EDA, Principal Investigator — Assiut University Hospitals
Locations (2):
- Assiut university hospitals, Asyut, Egypt
- Leeds teaching hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom